CLINICAL TRIAL: NCT03512171
Title: Dopaminergic Neuromodulation of Decision Making in Young and Middle-Aged Adults
Brief Title: Decision Making Study in Young and Middle-Aged Adults: Part II
Acronym: DND
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, David Zald, Cornelius Vanderbilt Professor of Psychology and Professor of Psychiatry, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 151088; AG043458 (Other Grant/Funding Number: MINH)
Record Dates: First submitted 2018-04-06; First posted 2018-04-30 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Dextroamphetamine

STUDY DESIGN:
Intervention Model Description: All subjects receive the same diagnositc intervention, with counterbalanced order
Who Masked: Participant, Investigator
Masking Description: The participant and the research analyst running their session are both blind, however a PET tech is unmasked who monitors the participant for any adverse reactions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Amphetamine (Experimental): One oral dose of dextroamphetamine (0.43 mg/kg) up to a maximum dose of 45mg. The dose is administered in 10mg and 2.5mg capsules prepared by the Vanderbilt Investigational Drug Services (IDS). Note: We are not testing the effect of dextro-amphetamine on a symptom. Rather it is part of the diagnostic intervention that is used to measure dopamine release assessed as the decline in [18F]fallypride binding relative to baseline.
  Interventions: Drug: Dextroamphetamine; Diagnostic Test: [18F]Fallypride
- Placebo (Placebo Comparator): One oral placebo dose, with capsules prepared by the Vanderbilt Investigational Drug Services (IDS). This provides the baseline against which dopamine release is measured.
  Interventions: Drug: Placebo; Diagnostic Test: [18F]Fallypride
- [18F]-FE-PE2I (Experimental): [18F]-FE-PE2I is a radioligand for measuring dopamine transporters with positron emission tomography (PET). All participants complete this arm. The arm does not include administration of amphetamine or placebo.
  Interventions: Diagnostic Test: [18F]-FE-PE2I

INTERVENTIONS:
Drug: Dextroamphetamine — One oral dose of dextroamphetamine (0.43mg/kg). The amphetamine is given in order to induce the release of their own dopamine for study with positron emission tomography (PET).
  Other Names: d-amphetamine
  Arms: Amphetamine
Drug: Placebo — One oral dose of placebo to estimate D2 receptor levels at baseline with PET imaging (necessary to calculate dopamine release in the amphetamine condition).
  Arms: Placebo
Diagnostic Test: [18F]Fallypride — Radioligand for measuring dopamine D2 receptors with positron emission tomography (PET)
  Other Names: [18F]Fallypride positron emission tomography
  Arms: Amphetamine; Placebo
Diagnostic Test: [18F]-FE-PE2I — Radioligand for measuring dopamine transporters with positron emission tomography (PET)
  Other Names: [18F]-FE-PE2I positron emission tomography
  Arms: [18F]-FE-PE2I

SUMMARY:
Financial decisions are made during pre-retirement age that can influence financial well-being for the rest of an individual's life. This proposal aims to construct a more comprehensive model of the specific psychological and neural mechanisms that support financial decisions in young adulthood and late middle age. In Part 1 of this study (covered in Institutional Review Board (IRB) # 141812), middle-age and young adults complete basic cognitive, motivational, and decision making tasks and are studied with functional magnetic resonance imaging (fMRI) to determine the relation between neural circuit activation and individual and age-related differences in decision making. In part II of the study, aspects of dopamine functioning are studied using positron emission tomography (PET) scanning to determine whether individual differences in dopamine functions are related to the decision-making and fMRI measures collected in Part 1 of the study. Dopamine measures include baseline D2 receptor availability, amphetamine induced dopamine release and dopamine transporter (DAT) levels, which provides a more comprehensive evaluation of dopamine functions than in prior studies linking individual differences in dopamine to behavioral, cognitive or decision-making traits.

DETAILED DESCRIPTION:
The study involves 4 sessions: 1) Informed Consent; 2) Oral d-amphetamine with Fallypride PET; 3) Placebo with Fallypride PET; and 4) PE2I PET. The oral amphetamine/placebo conditions utilize a double-blind counterbalanced design. The 3 PET sessions will be conducted within a 6 week window, and whenever possible within a 2 week time period.

1) Informed consent session: Informed consent will be obtained by Dr. Zald or approved study personnel after inclusion and exclusion criteria have been reviewed. Participants are screen for inclusion/exclusion as part of a separate IRB protocol (Vanderbilt IRB protocol #141812). After the consent processes is completed, participants will also complete the Tests of Vigilance and Attention (TOVA: http://www.tovatest.com/), which assesses attention abilities and motor impulsivity.

2 & 3) D-amphetamine/Placebo Fallypride PET Sessions

Participants complete two [18F]fallypride PET sessions, each lasting approximately 7 hours. Scan sessions will all start in the afternoon. Subjects will be instructed to have a moderate lunch with no more than a single cup of coffee or tea before coming to the PET center. If the scan is not expected to start until after 5 PM, a light snack may also be eaten. After determination of blood pressure, respirations, pulse, temperature, an intravenous line will be placed in the forearm, the subject will complete ratings of their mood (using the and PANAS and the Amphetamine Interview Schedule administered on a laptop computer), and participants will have a brief neurological exam conducted by one of the study MDs. An initial blood sample for genotyping or estradiol levels (women only) will be acquired.

The subject will then receive a 0.43 mg/kg oral dose of d-amphetamine or placebo. The investigational pharmacy will prepare capsules with 10 mg, and 2.5 mg with dosing rounded to the nearest 2.5 mgs (for instance an individual weighing 80 kg would be rounded up to a 35 mg dose). The drug dose and placebo, will be placed by the pharmacist in identical containers, labeled with the subject's ID and scan day number. A sealed envelope indicating whether the dose is d-amphetamine or placebo will be included in case there is a need to break the blinding. The study physician, can quickly access this information if there is appearance of an adverse drug effect. Otherwise the study physician and experimenters who have contact with the participant will remain blind until the participant has completed their second PET scan. If a participant has an adverse event that necessitates any medication, or other intervention, the blind will be broken to the participant.

Subjects will have blood pressure and pulse determinations every 30 minutes for the first 2.5 hours, prior to the start of PET scanning (around 175 minutes post-administration) and every 60-70 minutes thereafter until the subject's blood is in the normotensive range. In the event that the participant's blood pressure exceeds 180 mm Hg systolic, blood pressure will be measured every 15 minutes until it shows evidence of reducing (at least a 5 mm Hg decline). In the unlikely event that a subject's blood pressure should rise to greater than 200 mm Hg systolic B.P. for over 30 minutes, the patient may be treated with intravenous nitroprusside at the discretion of the study MD (see risk section below for specific details). We note that in our multi-year experience working with oral amphetamine, we have never required such an intervention.

After .5, 1, 1.25, 1.5, 2, 3, hours post-dAMPH/placebo administration and after the first two PET scans, approximately 4 and 5 hours subjects will complete ratings of mood (with selected items from the Amphetamine Interview Schedule and PANAS) and the DEQ (which asks them to rate whether they feel the drug, feel high, like the drug, or want more of the drug). Subjects will make their ratings on a laptop computer.

Cognitive Assessments: To further assess the cognitive specificity of dAMPH effects on cognition, participants will complete a battery of cognitive measures under placebo and drug. After the 60-minute post-administration blood pressure, mood ratings and blood draw, participants will begin performing the cognitive assessments tasks. Testing will include measures of speed of processing [WAIS-III Digit Symbol Coding and Symbol Search [115]], a measure of the speed of verbal associations [Controlled Oral Word Association Test [116]], and a measure of motor speed [finger tapping [151]] and a measure of working memory (2-back task). All tasks are included based on literature indicating that these functions are modulated by DA (e.g., [124,125]), with the tasks starting immediately following the amphetamine. The precise order of these tasks will vary, with brief tasks occurring during the 60-75 post-administration period, and the other tasks occurring following the 90 minute blood pressure and mood ratings.

Decision Making and Reward Learning Tasks. A 15-minute behavioral variant of the EEfRT task (which requires participants to make decisions about expending effort for rewards) will be performed starting 75 minutes after drug administration. In approximately half the trials the trial will terminate immediately after the decision phase, skipping both the effort expenditure and feedback phase. This approach allows us to complete significantly more decision trials during the 15 minute window.

Participants will also complete a two-stage reward learning paradigm that follows the procedures by Daw et al. (2011). On each trial, participants make an initial choice between two options labeled by Tibetan characters that lead probabilistically to either of two, second-stage "states," represented by different colors (see Figure 2). Each first stage choice is associated with one of the second stage states, and leads there 70% of the time. In turn, each of the second-stage states demanded another choice between another pair of options labeled by Tibetan characters. Each second-stage option was associated with a different probability of delivering a monetary reward (versus nothing) when chosen. To encourage participants to continue learning throughout the task, the chances of payoff associated with the four second-stage options is changed slowly and independently throughout the task, according to Gaussian random walks. In each stage participants have 2s to make a choice. Inter-stimuli and inter-trial intervals are 500ms and 300ms, respectively, and monetary reward is presented for 500ms. The task will take approximately 20 minutes to complete.

Spontaneous Eye Blinks: During portions of the study procedure participants may be asked to wear eye tracking goggles capable of recording spontaneous eye blinks. If participants cannot wear the goggles comfortably (primarily due to interactions with prescription glasses), will not be asked to wear the goggles.

Post administration blood draws: 4 blood draws (3 ml each) are taken to measure plasma amphetamine levels. These are collected at 30, 60, 90, and 175 minutes post-amphetamine. In order to avoid a different blood draw schedule, blood draws will additionally be made on the placebo day and will be discarded using appropriate hazardous biospecimen procedures. The lab will receive a sealed form that indicates whether to analyze or discard the samples.

PET scanning and fallypride administration: Scanning will be accomplished with a GE Discovery STE PET/CT scanner. 5 mCi of [18F]fallypride (specific activity > 3,000 Ci/mmol) will be injected, and subjects will be scanned for 3.5 hours (with two 15 minute breaks) to allow estimates of both striatal and extrastriatal binding potential. Dots are placed on the subject's forehead and cheeks for periodic visual checks of alignment throughout the scan period, and for repositioning after breaks. Three CT scans will also be collected during each session for attenuation correction. Blood pressure will be taken during each break and mood ratings will be taken during each break. During the second break participants will be given a high fat meal to help improve elimination of the radioisotope. Participants will also be given fluids to drink and asked to void their bladder.

At the conclusion of each PET scan on drug and placebo day, vital signs-blood pressure, pulse, temperature and respirations - will be measured, a brief motor neurological examination performed, and an additional 3.5 ml of blood drawn for a CBC and a comprehensive metabolic panel (CMP). If neurological exam and vital signs are normal the participants will be released from the study. In the unlikely event that they are not normal, the participant will be asked to stay under medical supervision in the VUMC (in one of the rooms in the PET center) until these measures have normalized. At the time of release participants will be given instructions to drink fluids and void their bladder at least once every two hours for up to 6 hours after the time of the start of the PET session.

4) FE-PE2I PET Session: Participants complete one [18F]FE-PE2I PET session lasting approximately 2 hours. Subjects will be instructed to not eat or drink coffee within 2 hours of the scheduled appointment. After determination of blood pressure, respirations, pulse, temperature, an intravenous line will be placed in the forearm, and a 3.5 ml blood sample for CBC and CMP will be drawn.

5 mCi of [18F]FE-PE2I (specific activity > NLT 457Ci/mmol) will be injected, and subjects will be scanned for 1 hour. Dots are placed on the subject's forehead and cheeks for periodic visual checks of alignment throughout the scan period. One CT scan will also be collected for attenuation correction.

At the conclusion of the PET scan, vital signs-blood pressure, pulse, temperature and respirations will be measured, and an additional 3.5 ml of blood will be drawn for a CBC CMP. Participants will be given a high fat snack or meal to help improve elimination of the radioisotope. They will also be given fluids to drink and asked to void their bladder. Participants will be given a neurological exam, and if both neurological exam and vital signs are normal, the participants will be released from the study. In the unlikely event that the neurological exam and vital signs are not normal, the participant will be asked to stay under medical supervision in the VUMC (in one of the rooms in the PET center) until these measures have normalized. At the time of release participants will be given instructions to drink fluids and void their bladder at least once every two hours for up to 6 hours after the time of the start of the PET session.

Specific procedures for female subjects of child-bearing potential: Premenopausal without hysterectomy or similar procedure, will need to have an additional blood draw within 48 hours prior to each PET session to rule out pregnancy (blood drawers will typically be scheduled within 36 hours preceding the planned time of radioisotope administration). Women who are premenopausal will be only studied within the first 10 days of their menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

Medically, psychiatrically and neurologically healthy individuals between the 20-30 or 50-65 years of age. Subjects must be able to give informed consent, have an estimated intelligence quotient of greater than 80, and be a fluent English speaker.

Exclusion Criteria:

1. Any condition which would interfere with or be a risk for MRI ( e.g. extreme obesity, claustrophobia, cochlear implant, metal fragments in eyes, cardiac pacemaker, neural stimulator, metallic body inclusions or other metal implanted in the body, facial tattoos with iron pigment). Difficulty lying on one's back and claustrophobia are also exclusions.
2. History of major psychiatric illness (including recurrent major depressive episodes or a depressive episode in the past 10 years, any anxiety disorders in the last 10 years, any history of bipolar disorder or psychotic disorder, a history of substance dependence (or substance abuse lasting more than 2 years), or any eating disorder in which symptoms persisted for more than two years
3. Current tobacco use, alcohol intake greater than 8 ounces of whiskey or equivalent per week, use of any psychotropic medication for the past 6 months (other than occasional use of benzodiazepines for sleep), psychostimulants taken more than 5 times in the subject's life, current marijuana use 4 Neurological illness (other than headache or strictly peripheral nerve disturbance), or head trauma (including more than 2 concussions)

5) Significant untreated or unregulated major medical condition deemed likely to influence cognitive functioning, dopaminergic functioning or neuroimaging measures. Diabetes is an exclusion even if well-controlled.

6) History of Syncope during blood draws 7) Anemia or hematocrit < 34. 8) Participation in any research studies in the past year that involved radiation, or exposure to radiation on a routine basis due to their occupation.

9) High blood pressure (Systolic B.P. > 150 in participants under the age of 61, or > 145 in subjects > 61 years of age). Diagnosis of labile hypertension. Abnormal EKG indicating potential cardiac risk under conditions of increased blood pressure.

10) Current pregnancy or lactation or plans to become pregnant during the study timeframe.

As part of the screening process in protocol # 141812, participants are initially screened with a brief telephone interview to determine if they meet medical, psychiatric and neurological criteria (all information screened is included in attached screening form). Participants are not consented until after completion of the brief health interview (a waiver of consent is in place in order to perform the initial telephone screening). After being consented participants complete a medical history and physical exam with one of the study MD's. They also complete a psychiatric interview (SCID-IV or V) with one of the trained psychology research assistants or Dr. Zald, and finally an EKG is completed. Participants are not enrolled in the present phase of the study until all exclusion criteria are assessed and they are withdrawn from the study if new information arises that would alter the conclusion regarding any of the inclusion/exclusion criteria after enrollment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Total number of participants planned is 60 broken into 30 females and 30 males.
Enrollment: 65 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Dopamine D2 receptor availability (binding potential) | 3- 6.5 hours
  D2 receptor availability is measured using positron emission tomography (PET) and the D2/D3 receptor radioligand [18F] fallypride. Contrast between receptor availability after amphetamine versus placebo forms the primary measure of dopamine release induced by amphetamine.

SECONDARY OUTCOMES:
Quantification of Dopamine Transporter Levels | 0 - 2 hours
  Dopamine transporter levels will be quantified with [18F]-FE-PE2I.
Decision Making Task 1 | 1-3 hours
  Effort Expenditure for Reward Task
Decision Making Task 2 | 1-3 hours
  Two-stage reward learning paradigm that follows the procedures by Daw et al. (2011)
Cognitive Task 1 (processing speed) | 1 - 2 hours
  WAIS-III Digit Symbol Coding and Symbol Search (aggregate score)
Cognitive Task 2 (verbal fluency) | 1 - 2 hours
  Controlled Oral Word Association Test
Cognitive Task 3 | 1 - 2 hours
  N-back task Working Memory Task (2-back & 3-back)
Motor Task 1 | 1 - 2 hours
  Finger Tapping Speed
Change in Spontaneous Eye Blink Rate | 1-2 hours
  Eye Blink Rate is measured with an eye tracker for 10 minutes, on or off amphetamine

CONTACTS AND LOCATIONS:
Overall Officials: David Zald, Zald, Principal Investigator — Vanderbilt University
Locations (1):
- Zald Affective Neuroscience Lab- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li SC, Lindenberger U, Sikstrom S. Aging cognition: from neuromodulation to representation. Trends Cogn Sci. 2001 Nov 1;5(11):479-486. doi: 10.1016/s1364-6613(00)01769-1. PMID 11684480
- [Background] Braver TS, Barch DM. A theory of cognitive control, aging cognition, and neuromodulation. Neurosci Biobehav Rev. 2002 Nov;26(7):809-17. doi: 10.1016/s0149-7634(02)00067-2. PMID 12470692
- [Background] Kaasinen V, Rinne JO. Functional imaging studies of dopamine system and cognition in normal aging and Parkinson's disease. Neurosci Biobehav Rev. 2002 Nov;26(7):785-93. doi: 10.1016/s0149-7634(02)00065-9. PMID 12470690
- [Background] Buckholtz JW, Treadway MT, Cowan RL, Woodward ND, Li R, Ansari MS, Baldwin RM, Schwartzman AN, Shelby ES, Smith CE, Kessler RM, Zald DH. Dopaminergic network differences in human impulsivity. Science. 2010 Jul 30;329(5991):532. doi: 10.1126/science.1185778. PMID 20671181
- [Background] Buckholtz JW, Treadway MT, Cowan RL, Woodward ND, Benning SD, Li R, Ansari MS, Baldwin RM, Schwartzman AN, Shelby ES, Smith CE, Cole D, Kessler RM, Zald DH. Mesolimbic dopamine reward system hypersensitivity in individuals with psychopathic traits. Nat Neurosci. 2010 Apr;13(4):419-21. doi: 10.1038/nn.2510. Epub 2010 Mar 14. PMID 20228805
- [Background] Zald DH, Cowan RL, Riccardi P, Baldwin RM, Ansari MS, Li R, Shelby ES, Smith CE, McHugo M, Kessler RM. Midbrain dopamine receptor availability is inversely associated with novelty-seeking traits in humans. J Neurosci. 2008 Dec 31;28(53):14372-8. doi: 10.1523/JNEUROSCI.2423-08.2008. PMID 19118170
- [Background] Ashby FG, Isen AM, Turken AU. A neuropsychological theory of positive affect and its influence on cognition. Psychol Rev. 1999 Jul;106(3):529-50. doi: 10.1037/0033-295x.106.3.529. PMID 10467897
- [Background] Carstensen LL, Turan B, Scheibe S, Ram N, Ersner-Hershfield H, Samanez-Larkin GR, Brooks KP, Nesselroade JR. Emotional experience improves with age: evidence based on over 10 years of experience sampling. Psychol Aging. 2011 Mar;26(1):21-33. doi: 10.1037/a0021285. PMID 20973600
- [Background] Carstensen LL, Pasupathi M, Mayr U, Nesselroade JR. Emotional experience in everyday life across the adult life span. J Pers Soc Psychol. 2000 Oct;79(4):644-55. PMID 11045744
- [Background] Charles ST, Carstensen LL. Emotion regulation and aging. Gross JJ, editor. Handbook of Emotion Regulation. New York: Guilford Press; 2007. p. 307-20.
- [Background] Carstensen LL. The influence of a sense of time on human development. Science. 2006 Jun 30;312(5782):1913-5. doi: 10.1126/science.1127488. PMID 16809530
- [Background] Carstensen LL, Isaacowitz DM, Charles ST. Taking time seriously. A theory of socioemotional selectivity. Am Psychol. 1999 Mar;54(3):165-81. doi: 10.1037//0003-066x.54.3.165. PMID 10199217
- [Background] Samanez-Larkin GR, Carstensen LL. Socioemotional Functioning and the Aging Brain. Decety J, Cacioppo JT, editors. The Handbook of Social Neuroscience. Oxford University Press; 2011. p. 507-21.
- [Background] Backman L, Ginovart N, Dixon RA, Wahlin TB, Wahlin A, Halldin C, Farde L. Age-related cognitive deficits mediated by changes in the striatal dopamine system. Am J Psychiatry. 2000 Apr;157(4):635-7. doi: 10.1176/ajp.157.4.635. PMID 10739428
- [Background] Volkow ND, Ding YS, Fowler JS, Wang GJ, Logan J, Gatley SJ, Hitzemann R, Smith G, Fields SD, Gur R. Dopamine transporters decrease with age. J Nucl Med. 1996 Apr;37(4):554-9. PMID 8691238
- [Background] Wang GJ, Volkow ND, Logan J, Fowler JS, Schlyer D, MacGregor RR, Hitzemann RJ, Gur RC, Wolf AP. Evaluation of age-related changes in serotonin 5-HT2 and dopamine D2 receptor availability in healthy human subjects. Life Sci. 1995;56(14):PL249-53. doi: 10.1016/0024-3205(95)00066-f. PMID 7475891
- [Background] Volkow ND, Logan J, Fowler JS, Wang GJ, Gur RC, Wong C, Felder C, Gatley SJ, Ding YS, Hitzemann R, Pappas N. Association between age-related decline in brain dopamine activity and impairment in frontal and cingulate metabolism. Am J Psychiatry. 2000 Jan;157(1):75-80. doi: 10.1176/ajp.157.1.75. PMID 10618016
- [Background] Volkow ND, Wang GJ, Fowler JS, Logan J, Gatley SJ, MacGregor RR, Schlyer DJ, Hitzemann R, Wolf AP. Measuring age-related changes in dopamine D2 receptors with 11C-raclopride and 18F-N-methylspiroperidol. Psychiatry Res. 1996 May 31;67(1):11-6. doi: 10.1016/0925-4927(96)02809-0. PMID 8797238
- [Background] Volkow ND, Wang GJ, Fowler JS, Ding YS, Gur RC, Gatley J, Logan J, Moberg PJ, Hitzemann R, Smith G, Pappas N. Parallel loss of presynaptic and postsynaptic dopamine markers in normal aging. Ann Neurol. 1998 Jul;44(1):143-7. doi: 10.1002/ana.410440125. PMID 9667606
- [Background] Kessler RM. Imaging methods for evaluating brain function in man. Neurobiol Aging. 2003 May-Jun;24 Suppl 1:S21-35; discussion S37-9. doi: 10.1016/s0197-4580(03)00047-2. PMID 12829104
- [Background] Christian BT, Narayanan T, Shi B, Morris ED, Mantil J, Mukherjee J. Measuring the in vivo binding parameters of [18F]-fallypride in monkeys using a PET multiple-injection protocol. J Cereb Blood Flow Metab. 2004 Mar;24(3):309-22. doi: 10.1097/01.WCB.0000105020.93708.DD. PMID 15091112
- [Background] Christian BT, Narayanan TK, Shi B, Mukherjee J. Quantitation of striatal and extrastriatal D-2 dopamine receptors using PET imaging of [(18)F]fallypride in nonhuman primates. Synapse. 2000 Oct;38(1):71-9. doi: 10.1002/1098-2396(200010)38:13.0.CO;2-2. PMID 10941142
- [Background] Mukherjee J, Christian BT, Dunigan KA, Shi B, Narayanan TK, Satter M, Mantil J. Brain imaging of 18F-fallypride in normal volunteers: blood analysis, distribution, test-retest studies, and preliminary assessment of sensitivity to aging effects on dopamine D-2/D-3 receptors. Synapse. 2002 Dec 1;46(3):170-88. doi: 10.1002/syn.10128. PMID 12325044
- [Background] Mukherjee J, Yang ZY, Brown T, Lew R, Wernick M, Ouyang X, Yasillo N, Chen CT, Mintzer R, Cooper M. Preliminary assessment of extrastriatal dopamine D-2 receptor binding in the rodent and nonhuman primate brains using the high affinity radioligand, 18F-fallypride. Nucl Med Biol. 1999 Jul;26(5):519-27. doi: 10.1016/s0969-8051(99)00012-8. PMID 10473190
- [Background] Rieck RW, Ansari MS, Whetsell WO Jr, Deutch AY, Kessler RM. Distribution of dopamine D2-like receptors in the human thalamus: autoradiographic and PET studies. Neuropsychopharmacology. 2004 Feb;29(2):362-72. doi: 10.1038/sj.npp.1300336. PMID 14627996
- [Background] Li SC, Lindenberger U, Backman L. Dopaminergic modulation of cognition across the life span. Neurosci Biobehav Rev. 2010 Apr;34(5):625-30. doi: 10.1016/j.neubiorev.2010.02.003. Epub 2010 Feb 10. No abstract available. PMID 20152855
- [Background] Eppinger B, Hammerer D, Li SC. Neuromodulation of reward-based learning and decision making in human aging. Ann N Y Acad Sci. 2011 Oct;1235:1-17. doi: 10.1111/j.1749-6632.2011.06230.x. PMID 22023564
- [Background] Mohr PN, Li SC, Heekeren HR. Neuroeconomics and aging: neuromodulation of economic decision making in old age. Neurosci Biobehav Rev. 2010 Apr;34(5):678-88. doi: 10.1016/j.neubiorev.2009.05.010. Epub 2009 Jun 6. PMID 19501615
- [Background] Kaasinen V, Vilkman H, Hietala J, Nagren K, Helenius H, Olsson H, Farde L, Rinne J. Age-related dopamine D2/D3 receptor loss in extrastriatal regions of the human brain. Neurobiol Aging. 2000 Sep-Oct;21(5):683-8. doi: 10.1016/s0197-4580(00)00149-4. PMID 11016537
- [Background] West RL. An application of prefrontal cortex function theory to cognitive aging. Psychol Bull. 1996 Sep;120(2):272-92. doi: 10.1037/0033-2909.120.2.272. PMID 8831298
- [Background] Hicks LH, Birren JE. Aging, brain damage, and psychomotor slowing. Psychol Bull. 1970 Dec;74(6):377-96. doi: 10.1037/h0033064. No abstract available. PMID 4322220
- [Background] MacPherson SE, Phillips LH, Della Sala S. Age, executive function, and social decision making: a dorsolateral prefrontal theory of cognitive aging. Psychol Aging. 2002 Dec;17(4):598-609. PMID 12507357
- [Background] Rubin DC. Frontal-Striatal Circuits in Cognitive Aging: Evidence for Caudate Involvement. Aging, Neuropsychology, and Cognition. 1999;6(4):241-59.
- [Background] Salthouse TA. Why are there different age relations in cross-sectional and longitudinal comparisons of cognitive functioning? Curr Dir Psychol Sci. 2014 Aug 1;23(4):252-256. doi: 10.1177/0963721414535212. PMID 25382943
- [Background] Raz N. The Aging Brain Observed in Vivo: Differential Changes and Their Modifiers. Cabeza R, Nyberg L, Park D, editors. Cognitive neuroscience of aging: Linking cognitive and cerebral aging. Oxford University Press, New York, NY, US; 2005. p. 19-57.
- [Background] Wardle MC, Treadway MT, Mayo LM, Zald DH, de Wit H. Amping up effort: effects of d-amphetamine on human effort-based decision-making. J Neurosci. 2011 Nov 16;31(46):16597-602. doi: 10.1523/JNEUROSCI.4387-11.2011. PMID 22090487
- [Background] Treadway MT, Buckholtz JW, Cowan RL, Woodward ND, Li R, Ansari MS, Baldwin RM, Schwartzman AN, Kessler RM, Zald DH. Dopaminergic mechanisms of individual differences in human effort-based decision-making. J Neurosci. 2012 May 2;32(18):6170-6. doi: 10.1523/JNEUROSCI.6459-11.2012. PMID 22553023
- [Background] Samanez-Larkin GR, Mata R, Radu PT, Ballard IC, Carstensen LL, McClure SM. Age Differences in Striatal Delay Sensitivity during Intertemporal Choice in Healthy Adults. Front Neurosci. 2011 Nov 16;5:126. doi: 10.3389/fnins.2011.00126. eCollection 2011. PMID 22110424
- [Background] Riccardi P, Li R, Ansari MS, Zald D, Park S, Dawant B, Anderson S, Doop M, Woodward N, Schoenberg E, Schmidt D, Baldwin R, Kessler R. Amphetamine-induced displacement of [18F] fallypride in striatum and extrastriatal regions in humans. Neuropsychopharmacology. 2006 May;31(5):1016-26. doi: 10.1038/sj.npp.1300916. PMID 16237395
- [Background] Kessler RM, Mason NS, Jones C, Ansari MS, Manning RF, Price RR. [18F]N-allyl-5-fluoropropylepidepride (fallypride): radiation dosimetry, quantification of striatal and extrastriatal dopamine receptors in man. NeuroImage. 2000Aug.26;11:S32.
- [Background] Woodward ND, Zald DH, Ding Z, Riccardi P, Ansari MS, Baldwin RM, Cowan RL, Li R, Kessler RM. Cerebral morphology and dopamine D2/D3 receptor distribution in humans: a combined [18F]fallypride and voxel-based morphometry study. Neuroimage. 2009 May 15;46(1):31-8. doi: 10.1016/j.neuroimage.2009.01.049. Epub 2009 Feb 5. PMID 19457373
- [Background] Riccardi P, Baldwin R, Salomon R, Anderson S, Ansari MS, Li R, Dawant B, Bauernfeind A, Schmidt D, Kessler R. Estimation of baseline dopamine D2 receptor occupancy in striatum and extrastriatal regions in humans with positron emission tomography with [18F] fallypride. Biol Psychiatry. 2008 Jan 15;63(2):241-4. doi: 10.1016/j.biopsych.2007.03.022. Epub 2007 Jun 27. PMID 17586476
- [Background] Zald DH, Woodward ND, Cowan RL, Riccardi P, Ansari MS, Baldwin RM, Cowan RL, Smith CE, Hakyemez H, Li R, Kessler RM. The interrelationship of dopamine D2-like receptor availability in striatal and extrastriatal brain regions in healthy humans: a principal component analysis of [18F]fallypride binding. Neuroimage. 2010 May 15;51(1):53-62. doi: 10.1016/j.neuroimage.2010.02.006. Epub 2010 Feb 10. PMID 20149883
- [Background] Riccardi P, Zald D, Li R, Park S, Ansari MS, Dawant B, Anderson S, Woodward N, Schmidt D, Baldwin R, Kessler R. Sex differences in amphetamine-induced displacement of [(18)F]fallypride in striatal and extrastriatal regions: a PET study. Am J Psychiatry. 2006 Sep;163(9):1639-41. doi: 10.1176/ajp.2006.163.9.1639. PMID 16946193
- [Background] Stroop JE. Studies of interference in serial verbal reactions. J Exp Psychol Gen. 1935;:18643-62.
- [Background] Wechsler D. Wechsler Memory Scale, 3rd edition. San Antonio, TX: Psychological Corporation; 1997.
- [Background] Wechsler D. Wechsler Adult Intelligence Scale, 3rd Edition. San Antonio, TX: Psychological Corporation; 1997.
- [Background] Benton AL. Development of a multilingual aphasia battery. Progress and problems. J Neurol Sci. 1969 Jul-Aug;9(1):39-48. doi: 10.1016/0022-510x(69)90057-4. No abstract available. PMID 5820858
- [Background] Rogers R, Monsell S. Costs of a predictible switch between simple cognitive tasks. Journal of experimental psychology: General. 1995;124(2):207-31.
- [Background] Bryden PJ, Roy EA. A new method of administering the Grooved Pegboard Test: performance as a function of handedness and sex. Brain Cogn. 2005 Aug;58(3):258-68. doi: 10.1016/j.bandc.2004.12.004. PMID 15963376
- [Background] Ruff RM, Parker SB. Gender- and age-specific changes in motor speed and eye-hand coordination in adults: normative values for the Finger Tapping and Grooved Pegboard Tests. Percept Mot Skills. 1993 Jun;76(3 Pt 2):1219-30. doi: 10.2466/pms.1993.76.3c.1219. PMID 8337069
- [Background] Park DC, Schwarz N, editors. Cognitive aging: A primer. Psychology Press, New York, NY, US; 2000.
- [Background] Buckner RL. Memory and executive function in aging and AD: multiple factors that cause decline and reserve factors that compensate. Neuron. 2004 Sep 30;44(1):195-208. doi: 10.1016/j.neuron.2004.09.006. PMID 15450170
- [Background] Luciana M, Depue RA, Arbisi P, Leon A. Facilitation of working memory in humans by a d2 dopamine receptor agonist. J Cogn Neurosci. 1992 Winter;4(1):58-68. doi: 10.1162/jocn.1992.4.1.58. PMID 23967857
- [Background] Servan-Schreiber D, Bruno RM, Carter CS, Cohen JD. Dopamine and the mechanisms of cognition: Part I. A neural network model predicting dopamine effects on selective attention. Biol Psychiatry. 1998 May 15;43(10):713-22. doi: 10.1016/s0006-3223(97)00448-4. PMID 9606524
- [Background] Lipkus IM, Samsa G, Rimer BK. General performance on a numeracy scale among highly educated samples. Med Decis Making. 2001 Jan-Feb;21(1):37-44. doi: 10.1177/0272989X0102100105. PMID 11206945
- [Background] Moustafa AA, Cohen MX, Sherman SJ, Frank MJ. A role for dopamine in temporal decision making and reward maximization in parkinsonism. J Neurosci. 2008 Nov 19;28(47):12294-304. doi: 10.1523/JNEUROSCI.3116-08.2008. PMID 19020023
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Carver CS, White TL. Behavioral Inhibition, Behavioral Activation, and Affective Responses to Impending Reward and Punishment: The BIS/BAS Scales. Journal of Personality and Social Psychology. 1994;67(2):319-33.
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Background] Cloninger CR, Przybeck TR, Svrakic DM. The Tridimensional Personality Questionnaire: U.S. normative data. Psychol Rep. 1991 Dec;69(3 Pt 1):1047-57. doi: 10.2466/pr0.1991.69.3.1047. PMID 1784653
- [Background] Costa PT, McCrae RR. Normal personality assessment in clinical practice: The NEO Personality Inventory. Psychological Assessment. 1992Mar.;4(1):5-13.
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Carstensen LL, Lang FR. Future Time Perspective Scale. 1995.
- [Background] Knutson B, Samanez-Larkin GR, Kuhnen CM. Gain and loss learning differentially contribute to life financial outcomes. PLoS One. 2011;6(9):e24390. doi: 10.1371/journal.pone.0024390. Epub 2011 Sep 6. PMID 21915320
- [Background] Ersner-Hershfield H, Garton MT, Ballard K, Samanez-Larkin GR, Knutson B. Don't stop thinking about tomorrow: Individual differences in future self-continuity account for saving. Judgm Decis Mak. 2009 Jun 1;4(4):280-286. PMID 19774230
- [Background] Samanez-Larkin GR, Levens SM, Perry LM, Dougherty RF, Knutson B. Frontostriatal white matter integrity mediates adult age differences in probabilistic reward learning. J Neurosci. 2012 Apr 11;32(15):5333-7. doi: 10.1523/JNEUROSCI.5756-11.2012. PMID 22496578
- [Background] McClure SM, Laibson DI, Loewenstein G, Cohen JD. Separate neural systems value immediate and delayed monetary rewards. Science. 2004 Oct 15;306(5695):503-7. doi: 10.1126/science.1100907. PMID 15486304
- [Background] Treadway MT, Buckholtz JW, Schwartzman AN, Lambert WE, Zald DH. Worth the 'EEfRT'? The effort expenditure for rewards task as an objective measure of motivation and anhedonia. PLoS One. 2009 Aug 12;4(8):e6598. doi: 10.1371/journal.pone.0006598. PMID 19672310
- [Background] Platt ML, Huettel SA. Risky business: the neuroeconomics of decision making under uncertainty. Nat Neurosci. 2008 Apr;11(4):398-403. doi: 10.1038/nn2062. Epub 2008 Mar 26. PMID 18368046
- [Background] Cox RW. AFNI: software for analysis and visualization of functional magnetic resonance neuroimages. Comput Biomed Res. 1996 Jun;29(3):162-73. doi: 10.1006/cbmr.1996.0014. PMID 8812068

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT03512171/Prot_SAP_000.pdf